CLINICAL TRIAL: NCT06570460
Title: Long Term Effects of Oral Versus Transdermal Estrogen Replacement Therapy in Turner Syndrome - A Randomized Trial
Brief Title: Long Term Effects of Oral Versus Transdermal Estrogen Replacement Therapy in Turner Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AU2019TS2
Record Dates: First submitted 2019-12-04; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Turner Syndrome; Hypogonadism; Ovarian; Hormone Replacement Therapy; Estrogen Replacement Therapy; Estrogen Deficiency
Keywords: Turner syndrome; Hormone replacement therapy; Estrogen replacement therapy; Estrogen treatment; Long term side effects
MeSH Terms: conditions — Turner Syndrome; Hypogonadism | interventions — Estradiol; estradiol, estriol drug combination

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Masking Description: The patients with TS will be randomized to receive either oral (tablet) or transdermal (gel) estrogen replacement therapy. The study is not blinded, as both investigator and study participants know which medication, they are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral estrogen treatment (Active Comparator): Turner syndrome patients receiving oral estrogen treatment (Estrofem®)
  Interventions: Drug: 17-beta estradiol
- Transdermal estrogen treatment (Active Comparator): Turner syndrome patients receiving transdermal estrogen treatment (Divigel)
  Interventions: Drug: 17-beta estradiol
- Controls (No Intervention): Healthy age-matched controls receiving no treatment

INTERVENTIONS:
Drug: 17-beta estradiol — Treatment with orally administered estrogen for 6 months
  Other Names: Estrofem
  Arms: Oral estrogen treatment
Drug: 17-beta estradiol — Treatment with transdermally administered estrogen for 6 months
  Other Names: Divigel
  Arms: Transdermal estrogen treatment

SUMMARY:
This 14-month, phase IV, randomized controlled crossover trial aims to compare the effects of oral versus transdermal estrogen replacement therapy (ERT) in women with Turner syndrome (TS). The study's objectives are to clarify endocrine, metabolic, cardiovascular, and thromboembolic risk factors in TS after a wash-out period without estrogen (E2) treatment; compare the effects of oral versus transdermal (TD) ERT regimens; and examine the long-term effects of E2 administration via these two routes. The study involves 50 TS women aged 18-50 years and 50 control participants. TS participants are randomized to receive either oral or TD ERT for six months, followed by crossover to the alternate treatment for another six months. Prior to randomization, any existing ERT will be discontinued for a 1-month washout period. A second 1-month washout period will occur between the two 6-month treatment phases. Laboratory analyses and clinical investigations are performed after the first wash-out period, after the first six months of treatment, and after the last six months of treatment. We anticipate that this study may provide a basis for new and improved recommendations for sex hormone replacement therapy in TS.

DETAILED DESCRIPTION:
OBJECTIVES

1. Clarify endocrine, metabolic, cardiovascular and thromboembolic risk factors in Turner syndrome (TS) after a wash out period
2. Compare the effects of oral versus transdermal (TD) estrogen replacement therapy (ERT) in women with Turner syndrome
3. Examine long term effects of ERT via the two routes on endocrine, metabolic, cardiovascular, physiologic and thromboembolic risk endpoints

BACKGROUND Turner syndrome (TS) is a rare genetic condition affecting approximately 1 in 2,000 female births. A hallmark of TS is ovarian dysgenesis, leading to hypogonadism, premature ovarian failure, and infertility. Consequently, estrogen replacement therapy (ERT) is typically initiated around age 11-12 to induce puberty and continued until the average age of menopause (50-55 years), aiming for at least 42 years of adequate estrogen exposure.

Hypogonadism in TS is associated with various health complications. Importantly, estradiol (E2) replacement may mitigate these risks. Estrogen deficiency in TS affects cardiovascular health (hypertension, congenital cardiac disease, altered lipid profiles), metabolic function (diabetes, thyroid dysfunction, hepatic disorders, kidney disease, skeletal abnormalities), and is linked to neurocognitive and social challenges.

E2 can be administered orally or transdermally (TD), but it remains unclear whether either route offers specific advantages. There is ongoing debate regarding a potential increased thromboembolic risk in TS patients treated with oral E2. Epidemiological studies in postmenopausal women have reported an elevated thromboembolic risk associated with oral estrogen treatment, but to a lesser extent with TD administration. However, extrapolating data from postmenopausal women to TS patients is inappropriate, as women with TS receive estrogen as replacement therapy due to inadequate endogenous production. Furthermore, limited knowledge exists regarding the side effects of oral versus TD estrogen replacement therapy for TS patients.

MATERIALS AND METHODS

Study group:

Women aged 18-50 years with TS recruited primarily from the Department of Endocrinology at Aarhus University Hospital (n=50); 300 patients with TS are currently followed in the outpatient clinic. The investigators also have the opportunity to recruit from the Turner Association in Denmark, and finally the investigators do have contact with other outpatient clinics with TS patients in Denmark from where the investigators have previously recruited TS patients.

An age-matched control group of healthy women is included by advertisement (n=50).

Inclusion criteria:

For participants with TS:

* Diagnosis of TS regardless of karyotype
* Age 18-50 years
* Already receiving estrogen treatment

For healthy controls:

* Female
* Age 18-50 years
* Previously healthy
* Not receiving any medication
* Not using any form of contraceptive pills
* No mental or psychiatric disorders

Exclusion criteria:

* Active systemic chronic diseases
* Known or suspected breast cancer
* Known or suspected estradiol-dependent tumors (endometrial cancer or similar)
* Untreated endometrial hyperplasia
* Current or previous venous thromboembolism
* Acute or previous liver disease where liver enzymes are still elevated by a factor 3 or more
* Known hypersensitivity to the medications used
* Pregnancy
* Menopause (for the control group only)

Design:

A 14-month, phase IV, randomized controlled crossover study involving women with Turner Syndrome (TS) (n=50) and healthy, age-matched controls (n=50). TS participants are randomized to receive either oral or TD ERT for six months, followed by crossover to the alternate treatment for another six months. Prior to randomization, any existing ERT will be discontinued for a 1-month washout period. A second 1-month washout period will occur between the two 6-month treatment phases. Healthy controls will not receive any treatment. They will undergo a single set of assessments for comparison.

Laboratory analyses and clinical investigations will be conducted at the Department of Endocrinology and the associated Medical Research Unit at Aarhus University Hospital. These will include blood and urine sample collection, as well as specific clinical investigations. At baseline, both TS patients and healthy controls will undergo these assessments. Only TS patients will undergo follow-up assesments.

Clinical investigations:

* Insulin sensitivity assessment
* 24-hour blood pressure monitoring
* DEXA scan (Dual-Energy X-ray Absorptiometry)
* Bioelectrical impedance analysis (Multiplate)
* Comprehensive clinical examination
* Quality of life assessments using questionnaires
* SphygmoCor analysis
* VO2 max test using a stationary bike
* MRI of the thigh muscles to measure muscle cross-sectional area (CSA) and intramuscular fat content
* Isometric muscle strength testing and functional testing

STATISTICS Data will be summarized by treatment group and assessment time point. The investigators will use a mixed model with repeated measures analysis of variance (ANOVA) to compare the mean changes in each of the study variables between treatments over time. When appropriate, transformations or nonparametric methods will be used. All tests are two-tailed with a 5% level of significance. Data are presented as mean ± SE or median with CI for metrics not normally distributed.

PERSPECTIVES Patients with TS undergo hormone replacement therapy from puberty to menopause, spanning more than 40 years of treatment. To date, only two experimental studies have compared oral and TD ERT in TS, focusing solely on metabolic parameters and finding no differences between the two regimens. If the investigators' hypotheses are correct and if the side effects, including increased thromboembolic risk, are higher with oral than TD ERT, this project could be crucial for optimizing treatment, improving quality of life, and reducing morbidity and mortality in TS. The investigators aim for this study to provide a basis for new and improved national and international recommendations for ERT in TS patients and to contribute new knowledge about hormonal treatment for the general population as well.

ELIGIBILITY:
Inclusion criteria:

For participants with TS:

* Diagnosis of TS regardless of karyotype
* Age 18-50 years
* Already receiving estrogen treatment

For healthy controls:

* Female
* Age 18-50 years
* Previously healthy
* Not receiving any medication
* Not using any form of contraceptive pills
* No mental or psychiatric disorders

Exclusion criteria:

* Active systemic chronic diseases
* Known or suspected breast cancer
* Known or suspected estradiol-dependent tumors (endometrial cancer or similar)
* Untreated endometrial hyperplasia
* Current or previous venous thromboembolism
* Acute or previous liver disease where liver enzymes are still elevated by a factor 3 or more
* Known hypersensitivity to the medications used
* Pregnancy
* Menopause (for the control group only)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only patients with Turner syndrome can participate and age mathed healthy controls (women)
Enrollment: 50 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood test values | After 1 month of wash-out, 6 months of oral and six months of transdermal treatment
  Changes in blood test values of follicle stimulating hormone and luthenizing hormone from baseline
Blood test values | After 1 month of wash-out, 6 months of oral and six months of transdermal treatment
  Changes in blood test values of estradiol from baseline
Dual energy X-ray absorptiometry | After 6 months of oral and six months of transdermal treatment
  Changes in body composition and bone mineral density
Cardiovascular status | After 6 months of oral and six months of transdermal treatment
  Changes in 24-hour blood pressure measurements
Cardiovascular status | After 6 months of oral and six months of transdermal treatment
  Changes in arterial stiffness measured by SphygmoCor
Muscle quality (quadriceps femoris) | After 6 months of oral and six months of transdermal treatment
  MR scan of both quadriceps measuring muscle cross-sectional area (CSA) and fat content of the muscle. Maximal isometric muscle strength of both quadriceps (functional muscle tests). Muscle quality = maximum quadriceps strength measured in nM/muscle CSA.
Functional muscle tests | After 6 months of oral and six months of transdermal treatment
  Changes in maximal jumping height
Isometric muscle tests | After 6 months of oral and six months of transdermal treatment
  Changes in maximal isometric hand strength
Maximal oxygen uptake test (VO2 max) | After 6 months of oral and six months of transdermal treatment
  Changes in maximal oxygen uptake

SECONDARY OUTCOMES:
Self-reported health-related quality of life and functioning (SF-36) | After 6 months of oral and six months of transdermal treatment
  The Short Form 36 Health Survey is a self-reported quality of life questionnaire consisting of eight scaled scores. Each scale is transformed directly into a 0-100 scale, where a lower score indicates greater difficulty.
Self-reported quality of life (WHOQoL-Bref) | After 6 months of oral and six months of transdermal treatment
  The WHOQoL-Bref is a questionnaire where the participant's answers to 26 questions are used to create an overall quality of life profile. This profile includes scores for each dimension of the questionnaire: physical health, mental health, social relationships, and the participant's environment.
Subjective medication assesment | After 6 months of oral and six months of transdermal treatment
  Subjective assesment of the medication after 6 months of use

CONTACTS AND LOCATIONS:
Overall Officials: Claus H Gravholt, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stochholm K, Juul S, Juel K, Naeraa RW, Gravholt CH. Prevalence, incidence, diagnostic delay, and mortality in Turner syndrome. J Clin Endocrinol Metab. 2006 Oct;91(10):3897-902. doi: 10.1210/jc.2006-0558. Epub 2006 Jul 18. PMID 16849410
- [Background] Gravholt CH, Andersen NH, Conway GS, Dekkers OM, Geffner ME, Klein KO, Lin AE, Mauras N, Quigley CA, Rubin K, Sandberg DE, Sas TCJ, Silberbach M, Soderstrom-Anttila V, Stochholm K, van Alfen-van derVelden JA, Woelfle J, Backeljauw PF; International Turner Syndrome Consensus Group. Clinical practice guidelines for the care of girls and women with Turner syndrome: proceedings from the 2016 Cincinnati International Turner Syndrome Meeting. Eur J Endocrinol. 2017 Sep;177(3):G1-G70. doi: 10.1530/EJE-17-0430. PMID 28705803
- [Background] Hjerrild BE, Mortensen KH, Gravholt CH. Turner syndrome and clinical treatment. Br Med Bull. 2008;86:77-93. doi: 10.1093/bmb/ldn015. Epub 2008 Apr 9. PMID 18400842
- [Background] Gravholt CH, Landin-Wilhelmsen K, Stochholm K, Hjerrild BE, Ledet T, Djurhuus CB, Sylven L, Baandrup U, Kristensen BO, Christiansen JS. Clinical and epidemiological description of aortic dissection in Turner's syndrome. Cardiol Young. 2006 Oct;16(5):430-6. doi: 10.1017/S1047951106000928. PMID 16984695
- [Background] Mortensen KH, Andersen NH, Hjerrild BE, Horlyck A, Stochholm K, Hojbjerg Gravholt C. Carotid intima-media thickness is increased in Turner syndrome: multifactorial pathogenesis depending on age, blood pressure, cholesterol and oestrogen treatment. Clin Endocrinol (Oxf). 2012 Dec;77(6):844-51. doi: 10.1111/j.1365-2265.2012.04337.x. PMID 22233516
- [Background] Mauger C, Lancelot C, Roy A, Coutant R, Cantisano N, Le Gall D. Executive Functions in Children and Adolescents with Turner Syndrome: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2018 Jun;28(2):188-215. doi: 10.1007/s11065-018-9372-x. Epub 2018 Apr 27. PMID 29704077
- [Background] Hansen M. Female hormones: do they influence muscle and tendon protein metabolism? Proc Nutr Soc. 2018 Feb;77(1):32-41. doi: 10.1017/S0029665117001951. Epub 2017 Aug 29. PMID 28847313
- [Background] Greising SM, Baltgalvis KA, Lowe DA, Warren GL. Hormone therapy and skeletal muscle strength: a meta-analysis. J Gerontol A Biol Sci Med Sci. 2009 Oct;64(10):1071-81. doi: 10.1093/gerona/glp082. Epub 2009 Jun 26. PMID 19561145
- [Background] Canonico M, Plu-Bureau G, Lowe GD, Scarabin PY. Hormone replacement therapy and risk of venous thromboembolism in postmenopausal women: systematic review and meta-analysis. BMJ. 2008 May 31;336(7655):1227-31. doi: 10.1136/bmj.39555.441944.BE. Epub 2008 May 20. PMID 18495631
- [Background] Renoux C, Dell'aniello S, Garbe E, Suissa S. Transdermal and oral hormone replacement therapy and the risk of stroke: a nested case-control study. BMJ. 2010 Jun 3;340:c2519. doi: 10.1136/bmj.c2519. PMID 20525678
- [Background] Sweetland S, Beral V, Balkwill A, Liu B, Benson VS, Canonico M, Green J, Reeves GK; Million Women Study Collaborators. Venous thromboembolism risk in relation to use of different types of postmenopausal hormone therapy in a large prospective study. J Thromb Haemost. 2012 Nov;10(11):2277-86. doi: 10.1111/j.1538-7836.2012.04919.x. PMID 22963114
- [Background] Gravholt CH, Naeraa RW, Fisker S, Christiansen JS. Body composition and physical fitness are major determinants of the growth hormone-insulin-like growth factor axis aberrations in adult Turner's syndrome, with important modulations by treatment with 17 beta-estradiol. J Clin Endocrinol Metab. 1997 Aug;82(8):2570-7. doi: 10.1210/jcem.82.8.4127. PMID 9253336
- [Background] Taboada M, Santen R, Lima J, Hossain J, Singh R, Klein KO, Mauras N. Pharmacokinetics and pharmacodynamics of oral and transdermal 17beta estradiol in girls with Turner syndrome. J Clin Endocrinol Metab. 2011 Nov;96(11):3502-10. doi: 10.1210/jc.2011-1449. Epub 2011 Aug 31. PMID 21880799
- [Background] Torres-Santiago L, Mericq V, Taboada M, Unanue N, Klein KO, Singh R, Hossain J, Santen RJ, Ross JL, Mauras N. Metabolic effects of oral versus transdermal 17beta-estradiol (E(2)): a randomized clinical trial in girls with Turner syndrome. J Clin Endocrinol Metab. 2013 Jul;98(7):2716-24. doi: 10.1210/jc.2012-4243. Epub 2013 May 15. PMID 23678038
- [Background] Gravholt CH, Naeraa RW, Nyholm B, Gerdes LU, Christiansen E, Schmitz O, Christiansen JS. Glucose metabolism, lipid metabolism, and cardiovascular risk factors in adult Turner's syndrome. The impact of sex hormone replacement. Diabetes Care. 1998 Jul;21(7):1062-70. doi: 10.2337/diacare.21.7.1062. PMID 9653596
- [Background] Klein KO, Baron J, Colli MJ, McDonnell DP, Cutler GB Jr. Estrogen levels in childhood determined by an ultrasensitive recombinant cell bioassay. J Clin Invest. 1994 Dec;94(6):2475-80. doi: 10.1172/JCI117616. PMID 7989605
- [Background] Klein KO, Rosenfield RL, Santen RJ, Gawlik AM, Backeljauw PF, Gravholt CH, Sas TCJ, Mauras N. Estrogen Replacement in Turner Syndrome: Literature Review and Practical Considerations. J Clin Endocrinol Metab. 2018 May 1;103(5):1790-1803. doi: 10.1210/jc.2017-02183. PMID 29438552
- [Background] Berglund A, Stochholm K, Gravholt CH. The epidemiology of sex chromosome abnormalities. Am J Med Genet C Semin Med Genet. 2020 Jun;184(2):202-215. doi: 10.1002/ajmg.c.31805. Epub 2020 Jun 7. PMID 32506765